CLINICAL TRIAL: NCT05246241
Title: Preoperative Magnetic Resonance Imaging Abnormalities Predictive of Lumbar Herniation Recurrence Following Surgical Repair
Brief Title: Preoperative Magnetic Resonance Imaging Abnormalities Predictive of Lumbar Herniation Recurrence
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mehmet Kursat Karadag, Principal Investigator, Ataturk University
Other Study IDs: ATANEUROSURGERY-1
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: magnetic resonance imaging — Preoperative magnetic resonance imaging

SUMMARY:
There are currently no standard criteria for evaluating the risk of recurrent disk herniation following surgical repair. This study investigated the predictive values of five presurgical imaging parameters, paraspinal muscle quality, annular tear size, Modic changes, modified Pfirrmann's disc degeneration grade, and presence of sacralization or fusion.

Clinical status and MRI findings were evaluated before surgery and 4, 12, and 24 months post-surgery using a Visual Analog Scale (VAS), Oswestry Disability Index (ODI), and Short Form 36 (SF36).

ELIGIBILITY:
Inclusion Criteria:

* first operation for a single-level lumbar disk herniation
* no concurrent spinal pathology such as stenosis, spondylolisthesis, or deformity
* complete data on clinical and radiological parameters

Exclusion Criteria:

* the operation was for multi-level pathologies
* recurrent surgery
* exhibited concurrent spinal pathology
* was missing or incomplete clinical and radiological data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18-75 male and female single-level lumbar disk herniation
Sampling Method: Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Paraspinal muscle quality | Preoperative 1 month
  Simplified 3-tier classification
Annular tear size | Preoperative 1 month
  With computer as millimeter
Modic changes | Preoperative 1 month
  Modic classification
Disc degeneration grade | Preoperative 1 month
  modified Pfirrmann's classification
sacralization or fusion | Preoperative 1 month
  MRI findings

SECONDARY OUTCOMES:
Visual Analog Scale | 4, 12, and 24 months after surgery
  0-10 numerical scale (0=no pain, 10 =the worst pain)
Oswestry Disability Index (ODI) | 4, 12, and 24 months after surgery
  Oswestry Low Back Pain Disability Questionnaire
Short Form 36 (SF36) | 4, 12, and 24 months after surgery
  SF-36 Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ammerman J, Watters WC, Inzana JA, Carragee G, Groff MW. Closing the Treatment Gap for Lumbar Disc Herniation Patients with Large Annular Defects: A Systematic Review of Techniques and Outcomes in this High-risk Population. Cureus. 2019 May 7;11(5):e4613. doi: 10.7759/cureus.4613. PMID 31312540
- [Background] Parker SL, Mendenhall SK, Godil SS, Sivasubramanian P, Cahill K, Ziewacz J, McGirt MJ. Incidence of Low Back Pain After Lumbar Discectomy for Herniated Disc and Its Effect on Patient-reported Outcomes. Clin Orthop Relat Res. 2015 Jun;473(6):1988-99. doi: 10.1007/s11999-015-4193-1. PMID 25694267